CLINICAL TRIAL: NCT04744662
Title: A Phase 1b Multicenter, Randomized, Controlled, Multi-dose Study of the Safety and Tolerability of ONL1204 Ophthalmic Solution in Patients With Geographic Atrophy (GA) Associated With Age-related Macular Degeneration (AMD
Brief Title: ONL1204 Ophthalmic Solution in Patients With Geographic Atrophy Associated With Age-related Macular Degeneration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ONL Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONL1204-GA-001
Record Dates: First submitted 2020-11-13; First posted 2021-02-09 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Geographic Atrophy
MeSH Terms: conditions — Geographic Atrophy | interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: In this study patients will be enrolled and followed for 24 weeks (natural history phase) at which point they will be randomized to 1 of 2 doses of ONL1204 Ophthalmic Solution or sham. Weeks 24 to 48 make up the Treatment Phase. Patients will be on study for a total of 48 weeks.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment Group A (Experimental): ONL1204 Ophthalmic solution (dose A) administered by intravitreal injection
  Interventions: Drug: ONL1204 Ophthalmic solution
- Treatment Group B (Experimental): ONL1204 Ophthalmic solution (dose B) administered by intravitreal injection
  Interventions: Drug: ONL1204 Ophthalmic solution
- Treatment Group C (Sham Comparator): sham injection without penetrating the eye
  Interventions: Procedure: sham injection

INTERVENTIONS:
Drug: ONL1204 Ophthalmic solution — Liquid formulation administered by intravitreal (IVT) injection
  Arms: Treatment Group A; Treatment Group B
Procedure: sham injection — sham injection is done by touching the eye surface with a syringe without a needle
  Arms: Treatment Group C

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of intravitreal injection of ONL1204 Ophthalmic Solution in patients with geographic atrophy associated with AMD.

GA associated with AMD is one of the world's leading causes of visual disability. It is a progressive disease with no approved therapy to slow or arrest the process of continual photoreceptor and retinal epithelial (RPE) cell loss. A safe and effective therapy for GA will have vast societal benefits. ONL1204 is being developed for this purpose. ONL1204 is a first-in-class inhibitor of fragment apoptosis stimulator receptor-mediated cell death in development for to reduce rates of vision in patients with GA associated with AMD. ONL1204 has demonstrated protection of multiple retinal cell types in several preclinical models of acute ocular injury and the protection of RPE in AMD models. ONL1204 Ophthalmic Solution is currently in a Phase 1 clinical study in patients with macula-off retinal detachment to evaluate safety and tolerability of a multi-dose of ONL1204 Ophthalmic Solution. The study is ongoing and uses the same doses and route of administration as this Phase 1b study in patients with GA.

DETAILED DESCRIPTION:
In this study patients will be enrolled and followed for 24 weeks (natural history phase) at which point they will be randomized to 1 of 2 doses of ONL1204 Ophthalmic Solution or sham. Weeks 24 to 48 make up the Treatment Phase. Patients will be on study for a total of 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, ≥ 55 years old
* Able to give informed consent and attend study visits
* Bilateral GA secondary to AMD without choroidal neovascularization in either eye
* ETDRS BCVA 20/400 (Snellen equivalent) or better in both eyes
* GA ≥1 disc area (DA) (DA, 2.5 mm2)
* If GA in study eye is multifocal, at least one focal lesion must have a DA of ≥ 1.25 mm2
* Entire GA area must be visible within the standard FAF field of view
* Presence of banded or diffuse hyperautofluoresence adjacent to GA lesion in study eye
* Female subjects must be:
* Women of non-childbearing potential, or
* WOCBP with a negative pregnancy test at screening and willing to use permissible methods of contraception for the duration of the study
* Males with female partners of childbearing potential must agree to use permissible methods of contraception and agree to refrain from donating sperm for the duration of the study.

Exclusion Criteria:

* GA in either eye due to causes other than AMD
* Participation in other ophthalmic clinical trials or use of any other investigational drugs or devices in study eye or systemically for 6 months prior to enrollment, or anticipated participation in other ophthalmic clinical trials or use of any other investigational drugs or devices in study eye or systemically during the study period
* Intraocular inflammation in the study eye
* Ocular or periocular infection in the study eye
* Media opacity that would limit baseline visual acuity or clinical visualization of the retina at baseline
* Hyperautofluoresence adjacent to GA lesion in study eye that is focal only
* Previous IVT treatment, history of retinal surgery, or other retinal therapeutic procedures in the study eye
* Systemic immunosuppression that may interfere with retinal and cytokine expression including but not limited to glucocorticoids (eg, oral prednisone or dexamethasone); antimetabolites (eg, methotrexate, mycophenolate mofetil, and azathioprine); T-cell inhibitors (eg, cyclosporine, tacrolimus, sirolimus); alkylating agents (eg, cyclophosphamide and chlorambucil); and biologic agents (eg, tumor necrosis factor inhibitors, interferons, lymphocyte inhibitors, and interleukin inhibitors)
* Prior history of systemic use of pentosan polysulfate sodium (trade name Elmiron®)
* Any ocular or systemic condition that in the opinion of the Investigator makes the subject unsuitable treatment with an investigational agent or that would compromise the safety and efficacy assessments of the trial
* An unwillingness to elect to either a) use Age-related Eye Disease Study 2 (AREDS2) formula nutraceutical therapy for the duration of the study or b) choose not to use such therapy for the duration of the study

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity | up to 48 weeks
  ETDRS chart (number of letters read)
Intraocular pressure | up to 48 weeks
  Intraocular pressure recorded in mmHg
Slit lamp biomicroscopy | up to 48 weeks
  Slit lamp using US FDA clinical grading scale 0-4; 0=normal, 4=very severe changes)

CONTACTS AND LOCATIONS:
Overall Officials: Robyn Guymer, MD, Principal Investigator — Center for Eye Research Australia
Locations (8):
- Australia (6):
  - Chatswood Retina, Chatswood, New South Wales
  - Retina and Eye Consultants Hurtsville, Hurstville, New South Wales
  - Retinology Institute, Glen Iris, Victoria
  - Queensland Eye Institute, Melbourne, Victoria
  - Center for Eye Rearch Australia, Melbourne, Victoria
  - Sunshine Eye Surgeons, St Albans, Victoria
- New Zealand (2):
  - Eye Institute Limited, Remuera, Auckland
  - Southern Eye Specialists, Christchurch